CLINICAL TRIAL: NCT04285164
Title: Normative Values of the Berg Balance Scale and Timed Up and Go Test in Elderly Females
Brief Title: Normative Values of the Berg Balance Scale and Timed Up and Go Test
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/Lhr/20/2016 Amna Anwar
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Community Dwelling Older Adults
Keywords: falls; Frail Elders; balance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Falls are a significant public health concern for older adults; early identification of people at high risk for falling facilitates the provision of rehabilitation treatment to reduce future fall risk. Berg balance scale is a reliable, valid and widely used tool to measure balance. Normal values of BBS declines with increasing age above 70 at a rate of 0.75 points per year. Timed up and go test Assess mobility, balance, falls risk. Normative data on both these test for our population is not established. Therefore this study aimed at finding normal scores of both these in our community-dwelling elderly females. For this purpose, data will be calculated from community-dwelling elderly females. BBS and TUG would be performed on each subject meeting our inclusion criteria after their consent. Data will be recorded and analyzed using Statistical Package for the Social Sciences (SPSS) version 23. We will find the mean and standard deviation. Thus this study will provide normal reference values of BBS and TUG in our community

DETAILED DESCRIPTION:
Balance deficits in elderly adults can arise from the process of ageing, such as age-related changes associated with the sensory system (vestibular, visual, somatosensory) or diseases such as cerebrovascular accident, arthritis, peripheral neuropathies, or disuse due to immobility. Balance is maintained when all the forces acting on the body are balanced so that one's centre of gravity is controlled within the base of support in static postures, during movement, and when responding to external disturbances. Normative data are important when interpreting any balance tool. the knowledge that a person or group of people Have worse balance than a healthy person of the same age may assist the identification and effective management of balance problem.

The BBS is a performance-based measure consisting of 14 items and a maximum score of 56. Originally developed to assess balance in older adults, it was subsequently adopted as a falls-risk prediction tool for older adults (although studies have differed in the recommended cut off score for falls risk. The BBS consists of 14 functional tasks of increasing difficulty, each scored from 0 to 4 (0¼unable to perform the task; 4¼task performed independently). The maximum score of 56 indicates no identifiable balance difficulties.

The 'timed up and go' test (TUG) is a simple, quick and widely used clinical performance-based measure of lower extremity function, mobility and fall risk. The TUG has been studied in elderly populations Women) the test procedure for the TUG is relatively simple. Subjects are asked to stand up from a standard chair (seat height between 44 and 47 cm), walk a distance of 3 m (marked on the floor) at a comfortable pace, turn, walk back and sit down. Subjects are permitted to use routine walking aids and are instructed not to use their arms to stand up. No physical assistance is given. The time to complete the task is measured with a stopwatch. Timing commences on the command 'go' and stops when the subject's back is positioned against the back of the chair after sitting down.

Use of local normative data of the specific population is recommended for more meaningful interpretation of TUG result Therefore, the aim of this study was to identify the normative data of TUG test and berg balance scale among community-dwelling older adults.the research was conducted in 2014 on normative scores on berg balance scale declines after age 70 in healthy community-dwelling people. it was a systematic review. purpose of this study was to find What is the mean Berg Balance Scale score of healthy elderly people living in the community and how does it vary with age? Group of healthy community-dwelling people with a mean age of 70 years or greater that has undergone assessment using the Berg Balance Scale were included. Mean and standard deviations of Berg Balance Scale scores within cohorts of elderly people of known mean age were measured. The mean Berg Balance Scale scores ranged from 37 to 55 out of a possible maximum score of 56. Although participants aged around 70 years had very close to normal Berg Balance Scale scores, there was a significant decline in balance with age at a rate of 0.7 points on the 56-point Berg Balance Scale per year. It was concluded that Healthy community-dwelling elderly people have modest balance deficits, as measured by the Berg Balance Scale, although balance scores deteriorate and become more variable with age.

the study was conducted on 'Timed Up and Go' test: Age, gender and cognitive impairment stratified normative values of older adults' in 2017. The aim of this study was to establish 'Timed up and Go' test (TUG) normative data among community-dwelling older adults stratified based on cognitive status, gender and age groups. A total of 2084 community-dwelling older adults from wave I and II were recruited through a multistage random sampling method. TUG was performed using the standard protocol and scores were then stratified based on with and without mild cognitive impairment (MCI), gender and in 5-year age groups ranging from ages of the '60s to '80s. 529(16%) participants were identified to have MCI. descriptive analysis showed, participants with MCI, women and older in age took a longer time to complete TUG, as compared to men with MCI across all age groups with exceptions for some age groups. These results suggested that MCI needs to be taken into consideration when testing older adults using TUG, besides age and gender factors.

a study on "Berg balance scale" and "timed up and go" Discriminates between fallers and non-fallers, in people with Multiple S. Different cut-offs have been used for BBS. With a cut-off at >44; high specificity (90%) but low sensitivity (40%) were found. Using ≤55 as cut-off yielded high sensitivity (94%) but low specificity (32%).TUG has not shown discriminant ability. The aim was to examine discriminant validity for BBS and TUG; fallers vs. non-fallers and predictive properties using previously suggested cut-offs. Data from three samples of PwMS (n=220) with imbalance was used. Testing was conducted by experienced research physiotherapists. Participants were classified as fallers or non-fallers. Mann-Whitney U test and ROC were used. BBS median for fallers was 45 points (n:108) and for non-fallers 50 points (n:99). TUG median was 17.5 seconds (n=108) for fallers and 13.2 seconds (n=99) for non-fallers.BBs: Using >44 points as cut-off correctly identified 51% of the fallers and 37% of the non-fallers. Using ≤55 correctly identified 96% fallers and 15% non-fallers.TUG: A cut-off (19.34 seconds) was chosen by maximizing the sum of sensitivity and specificity resulting in sensitivity at 70% and specificity at 43%.

Susan W Muir et al. conducted a study in 2008 on Use of the Berg Balance Scale for Predicting Multiple Falls in Community-Dwelling Elderly People. it was A Prospective Study. The objective of this study was to examine the predictive validity of the Berg Balance Scale (BBS) for 3 types of outcomes-any fall (1 fall), multiple falls (2 falls), and injurious falls-by use of sensitivity, specificity, receiver operating characteristic (ROC) curves, area under the curve, and likelihood ratios. A sample of 210 community-dwelling older adults received a comprehensive geriatric assessment at baseline, which included the BBS to measure balance. Data on prospective falls were collected monthly for a year. They concluded that the use of the BBS as a dichotomous scale to identify people at high risk for falling should be discouraged because it fails to identify the majority of such people. The predictive validity of this scale for multiple falls is superior to that for other types of falls.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults aged 60-80 years
* only females
* Tolerance of balance and gait tasks without fatigue
* Able to walk independently Get in or out of a chair with or without assistive device
* Independent in self-care activities (eating, bathing, dressing)
* Able to follow instructions in able to perform the test required in the study

Exclusion Criteria:

* Elderly individuals with a history of recurrent falls
* Cognitive and neurological impairments
* History of transitory ischemic attack
* stroke Participants on a wheelchair

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — elderly females
Study Population: community-dwelling older adult females who are able to walk independently and can take self-care activities independently without any cognitive issues & any co-morbidity.
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | day 1
  Berg balance scale (BBS) is used for assessment of balance and fall risk, Higher scores on the BBS indicate greater independence and better ability to balance. In contrast, lower scores indicate a greater fall risk Items DESCRIPTION SCORE (0-4) Sitting to standing _____ Standing unsupported _____ Sitting unsupported _____ Standing to sitting _____ Transfers _____ Standing with eyes closed _____ Standing with feet together _____ Reaching forward with outstretched arm _____ Retrieving object from floor _____ Turning to look behind _____ Turning 360 degrees _____ Placing alternate foot on stool _____ Standing with one foot in front _____ Standing on one foot _____ TOTAL __/56
Timed up and go test | day 1
  Timed up and go test is used for the assessment of falls risk among elderly population. The Timed "Up and Go" (TUG) Test measures, in seconds, the time taken by an individual to stand up from a standard arm chair (approximate seat height of 46 cm, arm height 65 cm), walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair, and sit down.
  Normal healthy elderly usually complete the task in 10 seconds or less. Very frail or weak elderly with poor mobility may take 2 minutes or more.
  Clinical guide: <10 seconds = normal <20 seconds = good mobility, can go out alone, mobile without a gait aid <30 seconds = problems, cannot go outside alone, requires a gait aid A score of more than or equal to 14 seconds has been shown to indicate high risk of falls.

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Nawaz Malik, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang CY, Hsieh CL, Olson SL, Wang CH, Sheu CF, Liang CC. Psychometric properties of the Berg Balance Scale in a community-dwelling elderly resident population in Taiwan. J Formos Med Assoc. 2006 Dec;105(12):992-1000. doi: 10.1016/S0929-6646(09)60283-7. PMID 17185241
- [Background] Downs S, Marquez J, Chiarelli P. Normative scores on the Berg Balance Scale decline after age 70 years in healthy community-dwelling people: a systematic review. J Physiother. 2014 Jun;60(2):85-9. doi: 10.1016/j.jphys.2014.01.002. Epub 2014 Jun 13. PMID 24952835
- [Background] Patterson KK, Inness E, McIlroy WE, Mansfield A. A Retrospective Analysis of Post-Stroke Berg Balance Scale Scores: How Should Normal and At-Risk Scores Be Interpreted? Physiother Can. 2017;69(2):142-149. doi: 10.3138/ptc.2015-73. PMID 28539694
- [Background] Muir-Hunter SW, Clark J, McLean S, Pedlow S, Van Hemmen A, Montero Odasso M, Overend T. Identifying balance and fall risk in community-dwelling older women: the effect of executive function on postural control. Physiother Can. 2014 Spring;66(2):179-86. doi: 10.3138/ptc.2013-16. PMID 24799756
- [Background] Herman T, Giladi N, Hausdorff JM. Properties of the 'timed up and go' test: more than meets the eye. Gerontology. 2011;57(3):203-10. doi: 10.1159/000314963. Epub 2010 May 20. PMID 20484884
- [Background] Ibrahim A, Singh DKA, Shahar S. 'Timed Up and Go' test: Age, gender and cognitive impairment stratified normative values of older adults. PLoS One. 2017 Oct 3;12(10):e0185641. doi: 10.1371/journal.pone.0185641. eCollection 2017. PMID 28972994
- [Background] Carling A, Forsberg A, Nilsagård Y. "Berg Balance Scale" and "Timed Up and Go" discriminates between fallers and non-fallers, in people with MS. InSixth International Symposium on Gait and Balance in Multiple Sclerosis, Portland, OR, US, and September 9-10, 2016 2016.
- [Background] Muir SW, Berg K, Chesworth B, Speechley M. Use of the Berg Balance Scale for predicting multiple falls in community-dwelling elderly people: a prospective study. Phys Ther. 2008 Apr;88(4):449-59. doi: 10.2522/ptj.20070251. Epub 2008 Jan 24. PMID 18218822